CLINICAL TRIAL: NCT03568266
Title: Pharmacogenomics of Age-Specific, Asparaginase-Induced Hepatotoxicity in Patients With Acute Lymphoblastic Leukemia
Brief Title: Pharmacogenomics of Asparaginase Induced Hepatotoxicity
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9L-17-16; NCI-2018-00813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-17-16 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biospecimen Collection: Buccal swabs of prospective participants' saliva will be collected when participant achieves complete remission (during regular clinical visit) from their asparaginase treatment.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva

SUMMARY:
This pilot trial studies the impact of genetic information on developing liver damage caused by asparaginase in participants with newly diagnosed acute lymphoblastic leukemia. Testing saliva samples may help doctors find certain genetic markers that may predict whether participants will tolerate asparaginase, which is given as part of clinical care for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the association between the SOD2 rs4880 genotypes and asparaginase-induced hepatotoxicity in Hispanic patients.

II. To identify novel single nucleotide polymorphisms (SNPs) that are associated with asparaginase induced hepatotoxicity.

OUTLINE:

Participants' SOD2 rs4880 SNP genotype (based on saliva from buccal swabs) will be classified. Participants with the CC genotype will be compared to participants with the CT or TT genotype. Buccal swabs of prospective participants' saliva will be collected when participant achieves complete remission (during regular clinical visit). Retrospective participants will be identified through search of pharmacy records for those who received asparaginase within the last 5 years (2012-2017). Recurrent patients will be consented during their regular clinical visits and samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with acute lymphoblastic leukemia (ALL) - no prior treatment for ALL
* Receiving asparaginase as part of the primary treatment regimen
* Ability to understand and the willingness to sign a written informed consent
* For retrospective recruitment, those who have received asparaginase between 2012 and 2017; and are current patients of University of Southern California (USC)

Exclusion Criteria:

* Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed with Acute Lymphoblastic Leukemia (ALL) who are seen at USC facilities will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatotoxicity following treatment with asparaginase | Up to 6 months
  Hepatotoxicity per Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) and defined as > or = grade 3 of both aspartate aminotransferase (AST) and alanine aminotransferase (ALT), or > or = grade 3 bilirubin elevation.

CONTACTS AND LOCATIONS:
Overall Officials: Houda Alachkar, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States